CLINICAL TRIAL: NCT00993746
Title: Comparison of Onset of Action Between 2% Lidocaine Plus 0.5% Bupivacaine and 0.5% Bupivacaine in Brachial Plexus Anesthesia for Creation of Arteriovenous Fistula in ESRD Patient
Brief Title: 2% Lidocaine Plus 0.5% Bupivacaine Versus 0.5% Bupivacaine in Brachial Block for Creation of Arteriovenous (AV) Fistula
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Faculty of Medicine Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: si433/2009
Record Dates: First submitted 2009-09-27; First posted 2009-10-12 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2009-10

CONDITIONS: Infraclavicular Brachial Plexus Block
Keywords: Ultrasound guided infraclavicular brachial plexus block; Bupivacaine; Bupivacaine plus lidocaine; End stage renal disease; Arteriovenous fistula
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula | interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine plus lidocaine (Active Comparator): Group 1: bupivacaine 20 ml plus lidocaine 10 ml
  Interventions: Drug: Bupivacaine plus lidocaine
- Bupivacaine alone (Experimental): Group 2: bupivacaine 30 ml
  Interventions: Drug: Bupivacaine 30 ml

INTERVENTIONS:
Drug: Bupivacaine plus lidocaine — Bupivacaine 20 ml plus lidocaine 10 ml
  Other Names: Marcaine Xylocaine
  Arms: Bupivacaine plus lidocaine
Drug: Bupivacaine 30 ml — Bupivacaine 30 ml for ultrasound guided infraclavicular brachial plexus block
  Other Names: lidocaine, marcaine
  Arms: Bupivacaine alone

SUMMARY:
Will the technique of adding lidocaine to bupivacaine fasten the onset of bupivacaine alone for infraclavicular brachial plexus block in end-stage renal disease (ESRD) patient?

ELIGIBILITY:
Inclusion Criteria:

* ESRD patient for AVF procedure
* age >17 year
* BMI 20-35 kg/m2
* communicable

Exclusion Criteria:

* BMI > 35 kg/m2 BMI < 20 kg/m2 หรือ BW < 35 kg
* History of allergy to local anesthetic drugs
* Pre-operative neurological deficit, Neuromuscular disorder หรือ old CVA
* Psychiatric disorder
* Coagulation disorder
* Uncontrolled seizure
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
onset of sensory block | 24 hour

SECONDARY OUTCOMES:
onset of motor block | 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Orawan Pongrawewan, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Department of anesthesiology Siriraj Hospital Mahidol University, Bangkok, Thailand